CLINICAL TRIAL: NCT05776797
Title: AV Junction Ablation or Optimal Medical Treatment in PatiEnts With Cardiac Resynchronization Therapy and Permanent Atrial Fibrillation
Acronym: AMPER-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMPER-AF trial
Record Dates: First submitted 2023-02-10; First posted 2023-03-20 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: atrial fibrillation; atrioventricular junction ablation; biventricular pacing; heart rate control; cardiac resynchronization therapy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Patients fulfilling the enrolment criteria will be randomly (randomization with variable blocks of 4, 6, and 8 patients) allocated to intervention and control groups in a 1:1 ratio.
Masking Description: No masking will be used in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrioventricular junction ablation (AVJA) in patients with cardiac resynchronization therapy (CRT) (Experimental): Patients with cardiac resynchronization therapy (CRT) randomized in this arm will undergo atrioventricular junction ablation.
  Interventions: Procedure: Atrioventricular junction ablation in patients with cardiac resynchronization therapy (CRT)
- Optimal medication treatment in patients with cardiac resynchronization therapy (CRT) (Active Comparator): Patients with cardiac resynchronization therapy (CRT) randomized in this arm will receive optimal medication treatment.
  Interventions: Drug: Optimal medication treatment in patients with cardiac resynchronization therapy (CRT)

INTERVENTIONS:
Procedure: Atrioventricular junction ablation in patients with cardiac resynchronization therapy (CRT) — Ablation of the atrioventricular (AV) node is a procedure used to disrupt or break the electrical connection between the upper heart chambers (the atria) and the lower heart chambers (the ventricles).
  Arms: Atrioventricular junction ablation (AVJA) in patients with cardiac resynchronization therapy (CRT)
Drug: Optimal medication treatment in patients with cardiac resynchronization therapy (CRT) — Optimal medication therapy according to the prescription of the physician.
  Arms: Optimal medication treatment in patients with cardiac resynchronization therapy (CRT)

SUMMARY:
A study comparing atrioventricular junction ablation (AVJA) versus continued optimum medical rate control in patients with cardiac resynchronization therapy (CRT) and atrial fibrillation (AF) with suboptimal heart rate control on optimum medication.

DETAILED DESCRIPTION:
Patients fulfilling the enrolment criteria will be randomly (randomization with variable blocks of 4, 6, and 8 patients) allocated to intervention and control groups in a 1:1 ratio. AVJA will be done in patients belonging to the intervention group without undue delay after the randomization. The procedure will be repeated in case of recovery of AV nodal conduction during the trial.

CRT device will be programmed to a base rate of 70 bpm, hysteresis switched off, and rate response functions activated unless not tolerated by the patient. The triggered mode will be encouraged.

All patients will be regularly followed in outpatient clinics. Cross-over to the AVJA study arm will be considered and performed at any time during the trial at the discretion of the operators. This may particularly concern patients with clinical deterioration in terms of functional status, quality of life, systolic left ventricular function, and/or repeated hospitalization, and in whom biventricular pacing (BiVP%) <<100% could be suspected as a significant underlying factor.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with CRT using either a biventricular pacemaker/defibrillator or conduction system pacemaker (>6 months)
* Diagnosis of AF and classified as: permanent AF or recurrent persistent AF, requiring emergency visits and/or hospitalizations (at least one in recent year)
* Optimized HF medical treatment and rate control medication
* BiVP% + ventricular premature complex (VPC%) <99% and >85% during the minimum period of 1 month while already on optimum medical therapy (applicable only for patients with permanent AF)
* Age >18 and <85 years
* Signed informed consent

Exclusion Criteria:

* myocardial infarction (MI) or coronary artery bypass graft (CABG) <3 months
* Technical failure of the CRT system
* Intentional preference for spontaneous AV conduction
* Expected survival <1 year
* Other significant comorbidities and/or conditions that interfere with the proper conduction of the trial
* Dementia as assessed by mini-mental test (<23 points)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Heart failure (HF) events | 3 years
  The number of HF events will be observed.
36-Item Quality of Life (QoL) | 3 years
  QoL will be assessed using the 36-Item Quality of Life Questionnaire. QoL will be evaluated at 12, 24 and 36 months as a sum of points that are assigned to individual outcome measures, specifically to their change compared to the baseline.
  To score the SF-36, scales are standardized to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 3 years
  MLHFQ values will be recorded and evaluated at 12, 24 and 36 months. The questionnaire is comprised of 21 questions around several physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. The patient marks a 0 (zero) to 5 (five) scale to indicate the extent to which each itemized adversity of heart failure has prevented the patient from living as they wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
Dose of loop diuretics | 3 years
  Change in the dose of loop diuretics will be observed and recorded. This parameter will be evaluated at 12, 24 and 36 months as an increase or decrease of the dose compared to the baseline.
NYHA classification | 3 years
  Changes in the New York Heart Association classification (NYHA) will be observed. The NYHA classification values will be evaluated at 12, 24 and 36 months. The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain.

SECONDARY OUTCOMES:
All-cause death | 3 years
  Patient deaths from all causes will be observed, recorded and analysed.
Death from cardiovascular diseases (CV death) | 3 years
  Incidents of CV death will be observed, recorded and analysed.
Combined heart failure (HF) death and HF hospitalization | 3 years
  Incidents of combined heart failure (HF) death and HF hospitalization will be observed, recorded and analysed.
Time-averaged proportional change in NT-pro-Brain Natriuretic Peptide (NT-pro-BNP) | 3 years
  The time-averaged proportional change in NT-pro-BNP will be observed, recorded and analysed.
Days in the hospital because of heart failure (HF) | 3 years
  The number of days in the hospital because of heart failure (HF) will be recorded.
Time-averaged change in the NYHA class | 3 years
  The time-averaged change in the NYHA class will be observed, recorded and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Plášek, MD,PhD,FESC, Principal Investigator — University Hospital Ostrava
Locations (9):
- Czechia (9):
  - Hospital České Budějovice, České Budějovice, Jihočeský kraj
  - Regional Hospital Liberec, Liberec, Liberec Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Hospital Podlesí, Inc., Třinec, Moravian-Silesian Region
  - University Hospital Olomouc, Olomouc, Olomouc Region
  - St. Anne's University Hospital Brno, Brno, South Moravian
  - University Hospital Brno, Brno, South Moravian
  - Institute of Clinical and Experimental Medicine, Prague
  - Military University Hospital Prague, Prague

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Ousdigian KT, Borek PP, Koehler JL, Heywood JT, Ziegler PD, Wilkoff BL. The epidemic of inadequate biventricular pacing in patients with persistent or permanent atrial fibrillation and its association with mortality. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):370-6. doi: 10.1161/CIRCEP.113.001212. Epub 2014 May 17. PMID 24838004
- [Background] Koplan BA, Kaplan AJ, Weiner S, Jones PW, Seth M, Christman SA. Heart failure decompensation and all-cause mortality in relation to percent biventricular pacing in patients with heart failure: is a goal of 100% biventricular pacing necessary? J Am Coll Cardiol. 2009 Jan 27;53(4):355-60. doi: 10.1016/j.jacc.2008.09.043. PMID 19161886
- [Background] Ganesan AN, Brooks AG, Roberts-Thomson KC, Lau DH, Kalman JM, Sanders P. Role of AV nodal ablation in cardiac resynchronization in patients with coexistent atrial fibrillation and heart failure a systematic review. J Am Coll Cardiol. 2012 Feb 21;59(8):719-26. doi: 10.1016/j.jacc.2011.10.891. PMID 22340263
- [Background] Waranugraha Y, Rizal A, Setiawan D, Aziz IJ. The Benefit of Atrioventricular Junction Ablation for Permanent Atrial Fibrillation and Heart Failure Patients Receiving Cardiac Resynchronization Therapy: An Updated Systematic Review and Meta-analysis. Indian Pacing Electrophysiol J. 2021 Mar-Apr;21(2):101-111. doi: 10.1016/j.ipej.2020.12.005. Epub 2021 Feb 4. PMID 33548449
- [Background] Dong K, Shen WK, Powell BD, Dong YX, Rea RF, Friedman PA, Hodge DO, Wiste HJ, Webster T, Hayes DL, Cha YM. Atrioventricular nodal ablation predicts survival benefit in patients with atrial fibrillation receiving cardiac resynchronization therapy. Heart Rhythm. 2010 Sep;7(9):1240-5. doi: 10.1016/j.hrthm.2010.02.011. Epub 2010 Feb 13. PMID 20156595
- [Background] Levy WC, Mozaffarian D, Linker DT, Sutradhar SC, Anker SD, Cropp AB, Anand I, Maggioni A, Burton P, Sullivan MD, Pitt B, Poole-Wilson PA, Mann DL, Packer M. The Seattle Heart Failure Model: prediction of survival in heart failure. Circulation. 2006 Mar 21;113(11):1424-33. doi: 10.1161/CIRCULATIONAHA.105.584102. Epub 2006 Mar 13. PMID 16534009
- [Background] Bozkurt B, Coats AJS, Tsutsui H, Abdelhamid CM, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Michael Felker G, Filippatos G, Fiuzat M, Fonarow GC, Gomez-Mesa JE, Heidenreich P, Imamura T, Jankowska EA, Januzzi J, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, Seferovic P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal definition and classification of heart failure: a report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure: Endorsed by the Canadian Heart Failure Society, Heart Failure Association of India, Cardiac Society of Australia and New Zealand, and Chinese Heart Failure Association. Eur J Heart Fail. 2021 Mar;23(3):352-380. doi: 10.1002/ejhf.2115. Epub 2021 Mar 3. PMID 33605000
- [Background] Packer M. Development and Evolution of a Hierarchical Clinical Composite End Point for the Evaluation of Drugs and Devices for Acute and Chronic Heart Failure: A 20-Year Perspective. Circulation. 2016 Nov 22;134(21):1664-1678. doi: 10.1161/CIRCULATIONAHA.116.023538. PMID 27881506
- [Background] Hussain A, Misra A, Bozkurt B. Endpoints in Heart Failure Drug Development. Card Fail Rev. 2022 Jan 18;8:e01. doi: 10.15420/cfr.2021.13. eCollection 2022 Jan. PMID 35111335
- [Background] Huber A, Oldridge N, Hofer S. International SF-36 reference values in patients with ischemic heart disease. Qual Life Res. 2016 Nov;25(11):2787-2798. doi: 10.1007/s11136-016-1316-4. Epub 2016 Jun 18. PMID 27318487